CLINICAL TRIAL: NCT06634108
Title: Cardiovascular Genistein Therapy for Heart Failure Inflammation
Brief Title: Genistein in trAnSthyretin recePtor Amyloid caRdiomyopathy
Acronym: GASPAR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Greenstone Biosciences (Unknown); Stanford University (Other)
Responsible Party: Principal Investigator, Mark Chandy, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13179
Record Dates: First submitted 2024-05-29; First posted 2024-10-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Amyloid Cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Genistein

STUDY DESIGN:
Intervention Model Description: Phase 1b/2a study to evaluate
  1. the safety of escalating doses of genistein
  2. the effects on cardiac function and exercise capacity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genistein Treatment and Washout (Experimental): The Investigators plan to recruit 40 heart failure participants, including 20 participants with heart failure with reduced ejection fraction (LVEF<40%) and 20 participants with transthyretin amyloid (ATTR) cardiomyopathy. After an initial telephone call to screen participants, the Investigators will invite qualified people for informed consent and a baseline fasting blood draw. Participants will receive escalating doses of genistein after their baseline fasting blood and stool sample collections. At baseline and again at 3 months, the Investigators will also perform transthoracic echocardiography and a 6-minute walk test.
  Interventions: Drug: Genistein

INTERVENTIONS:
Drug: Genistein — The genistein capsules are manufactured and obtained from MCS Formulas, and each capsule contains 250 mg genistein and 50 mg inulin. The genistein is certified to be 98% pure genistein by HPLC and is certified by Good Laboratory Practice (GLP). They will consume 250 mg of genistein BID (500 mg total) by mouth for the first 4 weeks before blood and stool samples are collected. Then, participants will take 500 mg of genistein BID (1000 mg total) for the next 4 weeks before collecting fasting blood and stool samples. Afterward, participants will take 750 mg of genistein BID (1500 mg total) for 4 weeks before collecting fasting blood and stool samples. Afterward, participants will have a washout for 6 weeks before returning for fasting blood and stool sample collection.

SUMMARY:
This Phase 1b/2a study aims to investigate the safety and efficacy of genistein in patients with Transthyretin (TTR) Amyloidosis. The focus is on its impact on inflammatory and cardiometabolic biomarkers, along with the effects on cardiac function and exercise capacity.

Blood samples will be collected at baseline, following each dose of genistein, and after a six-week placebo washout period. These samples will undergo extensive analyses, including profiling for inflammatory cytokines and novel molecular markers, and routine tests like CBC, Chem 7, LFT, HbA1c, NT-proBNP, CRP, troponin T, and serum TTR. RNA-seq analyses on peripheral blood mononuclear cells (PBMCs) and isolation of plasma exosomes for inflammatory biomarkers are also part of the protocol.

Following ESC/AHA guidelines, echocardiography will assess cardiac structure and function, focusing on the left and right ventricles and valvular function. Additionally, exercise capacity will be evaluated through a standardized 6-minute walk test, and NT-proBNP levels will be measured as a cardiac stress biomarker.

The trial will include an 18-week follow-up period post-enrolment, with the primary endpoint being the change in inflammatory markers from baseline to three months. Secondary endpoints are cardiac function and exercise capacity changes over the same timeframe. This study aims to provide significant insights into genistein's therapeutic potential for TTR Amyloidosis and its broader implications in managing heart failure.

Following ethical committee approval and written informed consent, the Investigators aim is to enroll 40 participants. This is an open-label study. Each patient will receive genistein by mouth: 250 mg twice a day for 4 weeks (500 mg total/day), 500 mg twice a day for 4 weeks (1000 mg total/day), and 750 mg twice a day (1500 mg total/day) for an additional 4 weeks. This will be followed by a 6-week washout period to conclude the study. An 18-month study is anticipated based on the average enrollment rates. Results from this study are expected to offer critical insights for future larger studies.

DETAILED DESCRIPTION:
BACKGROUND.

Heart Failure (HF) is a complex clinical syndrome when the heart cannot meet the metabolic demands of the body. HF is a growing health and economic burden in the United States. Between 2013 to 2017, there were over 1.2 million hospitalizations per year and costs of over $30 billion per year. The prognosis of HF is quite poor, with the number of deaths per year increasing from 275,000 in 2009 to 310,000 in 2014.

HF is caused by ischemic cardiomyopathy, valvular disease, and non-ischemic cardiomyopathy, which includes infiltrative cardiac disease such as amyloidosis. The link between inflammation and HF is well characterized and plays a significant role in heart failure. The immune system is activated in response to myocardial injury, decreased peripheral perfusion, or neurohormonal activation. Cytokines are released from inflammatory cells and destabilize cardiovascular function. When a cardiomyocyte is damaged by infarction or stretch from volume or pressure overload, the surrounding myocytes secrete inflammatory cytokines that further exacerbate HF.

Inflammatory cytokines serve as reliable indicators of HF severity, providing prognostic value and a means to assess the effectiveness of therapeutic interventions. A host of inflammatory cytokines, such as interleukin-6 (IL-6), interleukin-8 (IL-8), tumor necrosis factor-a (TNF-alpha), and interferon g (IFN-gamma), have been identified as key players in the pathogenesis of HF. Chronic HF management includes correcting the underlying cause, treating symptoms, and long-term pharmacological and device therapy. In the chronic setting, pharmacological interventions such as β-blockers, ACE inhibitors, aldosterone antagonists, and sodium-glucose cotransporter-2 inhibitors (SGLT2i) combined with implantable cardioverter-defibrillator (ICD) and cardiac resynchronization therapy (CRT) can markedly improve symptoms and survival.

GENISTEIN

Genistein, a soybean derivative, can potentially reduce inflammation and oxidative stress, as demonstrated in numerous preclinical models. It has been studied extensively and has no known adverse side effects. Moreover, it does not significantly interact with cardiac medications.

Genistein has emerged as an interesting compound due to its anti-inflammatory and antioxidant properties. Acting as an antagonist to cannabinoid receptor 1, genistein can influence several pathways implicated in the exacerbation of heart failure, primarily inflammation and oxidative stress. Evidence from preclinical models has highlighted genistein's capacity to modulate immune responses and alleviate oxidative stress, which are instrumental in the inflammatory processes underlying heart failure. Moreover, genistein has demonstrated cardio-protective effects in various in vitro and animal studies, suggesting a therapeutic potential that warrants further clinical exploration.

ATTR PATHOGENESIS

Transthyretin amyloid cardiomyopathy (ATTR-CM) is an often-overlooked form of amyloidosis that leads to restrictive cardiomyopathy and progressive heart failure. This condition predominantly affects the elderly and patients with hypertrophic cardiomyopathy. ATTR-CM results from the aggregation of misfolded transthyretin (TTR) proteins, which form amyloid fibrils that deposit in the cardiac tissue. These deposits can disrupt normal cardiac architecture and function, precipitating diastolic dysfunction and heart failure.

The misfolding and aggregation of TTR, a protein responsible for transporting thyroxine and retinol-binding protein, can be attributed to genetic mutations or age-related changes. genistein has been shown to bind and stabilize TTR, potentially inhibiting its misfolding and subsequent fibril formation. This stabilization presents a novel approach that could impede the progression of ATTR-CM.

STUDY RATIONALE

A notable pathogenic process associated with aging or mutation involves the misfolding of Transthyretin (TTR), leading to its aberrant assembly into amyloid. This misassembly causes conditions such as amyloidosis, familial amyloid neuropathy, and amyloid cardiomyopathy. Small molecules have been found to stabilize the native tetramer by binding to the thyroid hormone binding sites of TTR.

The current clinical trial is designed to address a pivotal gap in heart failure treatment by integrating genistein as an adjunct therapy alongside the standard of care, tafamidis. By targeting both the inflammatory mechanisms implicated in heart failure and the molecular pathogenesis of ATTR-CM, the study positions genistein as a potential modifier of disease progression.

Recognized for its commendable safety profile and the absence of reported major adverse side effects, genistein holds the potential to address ATTR-CM. The adjunctive use of genistein could enhance tafamidis therapy, offering a dual approach to stabilize TTR and mitigate inflammation. This study is poised to contribute significantly to the heart failure therapeutic landscape, potentially improving outcomes for patients with ATTR amyloid cardiomyopathy. By exploring genistein's role in conjunction with established therapies, this research may pave the way for novel, more effective treatment regimens for heart failure, particularly in those with or at risk for ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-80 years
* Heart failure with Reduced Ejection Fraction

  * ischemic or nonischemic etiology
  * LVEF <40% by echocardiography, MUGA, or MRI
* ATTR cardiomyopathy

  * any LVEF by echocardiography, MUGA, or MRI
* Stable optimally tolerated dosages of HF therapies for 3 months with no change in medical management regimen for at least 1 month
* NT-proBNP

  * for participants < 75 years old with NT-proBNP > 125 pg/mL
  * for participants > 75 years old with NT-proBNP > 450 pg/mL

Exclusion Criteria:

* Coronary intervention in the past 3 months
* Pregnancy
* Endometriosis
* Uterine fibroids
* Cancer:

  * including breast cancer
  * predisposition to cancer such as abnormal mammogram
  * family history
  * BRCA1 or BRCA2 positive
  * Patients on a vegan diet
* Patients taking supplements such as isoflavonoid, genistein, or resveratrol
* Ethanol abuse
* Men: >4 drinks on any day or more than 14 drinks per week
* Women: >3 drinks on any day or more than 7 drinks per week
* Liver dysfunction:

  * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3X ULN
  * total bilirubin greater than 1.5 times ULN
* hormone replacement therapy (HRT)
* thyroid supplement
* Renal dysfunction (eGFR less than 25 mL/min/1.73 m2)
* Uncontrolled diabetes (HgbA1c >10%)
* Coagulopathies
* Cytopenia:

  * leukocytopenia
  * hemoglobin < 9 mg/dl
  * platelets <100x103/mm3
* Any patients who had been hospitalized in the past 3 months for reasons other than heart failure
* NYHA Functional Class I or Functional Class IV symptoms.
* Acute bacterial or viral infectious disease, or acute exacerbation of a chronic infectious disease
* allergy to genistein or inulin
* allergy to perflutren dye used in contrast echocardiography

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  To assess the safety profile and effect of genistein on key inflammatory biomarkers in patients with heart failure, the following markers will be assessed using specified measurements:
  Interleukin-6 (IL-6): Measured using ELISA. Interleukin-8 (IL-8): Measured using ELISA. Tumor Necrosis Factor-alpha (TNF-α): Measured using ELISA. Interferon-gamma (IFN-γ): Measured using ELISA.
Cardiac markers | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  To assess the safety profile and effect of genistein on key cardiometabolic biomarkers in patients with heart failure, the following markers will be assessed using specified measurements:
  B-type Natriuretic Peptide (BNP): Measured using immunoassay. C-reactive Protein (CRP): Measured using immunoassay.
Complete metabolic profile | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  To assess the safety profile and effect of genistein on key cardiometabolic biomarkers in patients with heart failure, the following markers will be assessed using specified measurements:
  Hemoglobin A1C (HgA1C): Measured using standard laboratory methods. Complete Blood Count (CBC): Measured using automated hematology analyzer. Comprehensive Metabolic Panel (Chem 7): Measured using standard laboratory methods.
  Liver Function Tests (LFT): Measured using standard laboratory methods.

SECONDARY OUTCOMES:
The impact of genistein on exercise capacity | This parameters will be assessed at baseline (week 0) and after washout (week 18).
  Exercise capacity will be evaluated by 6-minute walk test, which will be performed by a blinded observer according to the standard protocol.
The impact of genistein on cardiac volume | This parameters will be assessed at baseline (week 0) and after washout (week 18).
  Cardiac size will be evaluated by echocardiography. The scans will assess left ventricle end-systolic- and end-diastolic volumes (LVESV and LVEDV).
The impact of genistein on cardiac mass | This parameters will be assessed at baseline (week 0) and after washout (week 18).
  Cardiac mass will be evaluated by echocardiography.
The impact of genistein on cardiac systolic function | This parameters will be assessed at baseline (week 0) and after washout (week 18).
  Echocardiography will evaluate cardiac function. The scans will assess global left ventricular systolic function, left ventricular ejection fraction (LVEF), and RV systolic function.
The impact of genistein on cardiac diastolic function | This parameters will be assessed at baseline (week 0) and after washout (week 18).
  Echocardiography will evaluate cardiac function. The scans will assess LV diastolic function by E lateral and medial velocity, E/e', LA volume, and TR velocity.
The impact of genistein on cardiac function using strain imaging | This parameters will be assessed at baseline (week 0) and after washout (week 18).
  Left ventricular function will be evaluated by radial and longitudinal global and segmental strain by two-dimensional speckle-tracking echocardiography. Right ventricular two-dimensional speckle tracking derived longitudinal strain analysis of the RV free wall averaged over three right ventricular free wall segments.

OTHER OUTCOMES:
Exploratory Blood Biomarkers | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  The Investigators will assess alterations in blood biomarkers through unbiased proteomics post-Genistein treatment and benchmark against baseline. The specific biomarkers and measurement tools are as follows:
  Proteomics Analysis:
  * Platform: OLink or RayBiotech proteomic profiling array.
  * Biomarkers: A comprehensive panel of proteins related to inflammation, oxidative stress, and cardiovascular health will be assessed.
  Examples of Biomarkers:
  * Cytokines: IL-6, IL-8, TNF-α, IFN-γ.
  * Acute Phase Proteins: CRP, Serum Amyloid A.
  * Growth Factors: VEGF, EGF.
  * Metabolic Proteins: Adiponectin, Leptin.
  Units of Measure:
  • The biomarkers will be measured in their respective units, typically in picograms per milliliter (pg/mL) or nanograms per milliliter (ng/mL).
Microbiome DNA sequencing | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  The effects of genistein on the microbiome will be studied by collecting stool samples at baseline, after each dose escalation, and after washout. Participant stool samples will have DNA sequencing to detect alternations in the microbial flora with genistein treatment.
  Units of Measure:
  The DNA sequencing analysis will identify genetic signatures of microbial flora.
Microbiome RNA sequencing | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  The effects of genistein on the microbiome will be studied by collecting stool samples at baseline, after each dose escalation, and after washout. Participant stool samples will have RNA sequencing to detect alternations in the microbial flora with genistein treatment.
  Units of Measure:
  The RNA sequencing dataset will be normalized to the baseline as a relative fold expression.
Microbiome: | These parameters will be assessed at baseline (week 0) and with each dose escalation (week 4, week 8, and week 12) and after washout (week 18).
  The effects of genistein on the microbiome will be studied by collecting stool samples at baseline, after each dose escalation, and after washout. Participant stool samples will have metabolomics to detect alternations in the microbial flora with genistein treatment.
  Units of Measure:
  The metabolome will be assessed with mass spectrometry for changes in microbial metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Mark JK Chandy, MD PhD, Principal Investigator — Lawson
Locations (1):
- London Regional Health Science Centre, London, Ontario, Canada